CLINICAL TRIAL: NCT01976481
Title: Serum 25-OH Vitamin D Modulation by Sunbed Use According to EU Guideline EN 60335-2-27
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: sunbed study
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2015-08

CONDITIONS: Skin Toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunbed (Experimental): sunbed exposure
  Interventions: Device: sunbed exposure
- Observation (No Intervention): only observation of subjects recruited after randomization

INTERVENTIONS:
Device: sunbed exposure — exposure to sunbed ultraviolet radiation
  Arms: Sunbed

SUMMARY:
Our study aims to clarify the impact of the use of a standard sunbed according to new EU guideline EN 60335-2-27 and possibly discount the positive effects of tanning beds. We plan to investigate the serum elevation of 25(OH)D under sunbed use, respecting the new recommendations for the exposure plan for different skin types according to EN 60335-2-27.

The use of a sunbed will be compared to a control group not using a sunbed in the observation period.

* Trial with medical device

DETAILED DESCRIPTION:
We will compare to baseline changes in serum vitamin D and health-related quality of life using a control group and an intervention group.

ELIGIBILITY:
Inclusion criteria: Probands intending to use a commercial sunbed :

1. Age 18 years or older
2. Regular use of commercial sunbeds
3. Oral and written informed consent

Exclusion criteria: 1. Skin type I according to Fitzpatrick according to EU guideline EN 60335-2-27 2. Sunbed use within the last three months 3. Use of vitamin D supplements or multivitamin supplements 4. Any medical condition which renders them unfit for sunbed use in the judgment of the investigator 5. Inability to provide oral and written consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Determination of number of patients with a relevant elevation of serum 25-hydroxyvitamin D levels of =10ug/L from the baseline | six months

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Hofbauer, Prof MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No